CLINICAL TRIAL: NCT05915234
Title: Analysis of the Effect of Different Cryotherapy Procedures on the Radial Puncture Site for Blood Gas Analysis Randomized Controlled Trial
Brief Title: Effect of Cryotherapy Modalities on Skin Temperature, Radial Artery Size and Flow Where Arterial Puncture Are Performed
Acronym: ECCRIOGAS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been postponed indefinitely. It is likely to be carried out in 2026-27
Sponsor: Julio Alberto Mateos Arroyo (Other)
Collaborators: Universidad Complutense de Madrid (Other); Hospital General Nuestra Señora del Prado (Other)
Responsible Party: Sponsor-Investigator, Julio Alberto Mateos Arroyo, Principal Investigator, Hospital General Nuestra Señora del Prado
Organization: Hospital General Nuestra Señora del Prado (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECCRIOGAS
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Temperature; Blood Flow Velocity; Radial Artery Size
Keywords: Cryotherapy; Skin temperature; Radial artery; Hemodynamics

STUDY DESIGN:
Intervention Model Description: Randomized experimental model in which 2 active cryotherapy interventions and a control are applied to all participants in a crossover single-blind design.
Who Masked: Participant
Masking Description: This study uses a single-blind masking. The 2 interventions and the comparator are contained in opaque bags, that prevents participants from having visual knowledge of the contents of the bags.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Order number 1: Ice-Peas-Control (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: crushed ice - frozen peas - control.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel
- Order number 2: Ice-Control-Peas (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: crushed ice - control - frozen peas.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel
- Order number 3: Peas-Ice-Control (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: frozen peas - crushed ice - control.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel
- Order number 4: Peas-Control-Ice (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: frozen peas - control - crushed ice.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel
- Order number 5: Control-Ice-Peas (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: control - crushed ice - frozen peas.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel
- Order number 6: Control-Peas-Ice (Experimental): Each subject will receive all interventions and the control and they will randomly assigned to a sequence order. In this arm the sequence order is: control - frozen peas - crushed ice.
  Interventions: Device: Crushed ice; Device: Frozen peas; Device: Room temperature gel

INTERVENTIONS:
Device: Crushed ice — Each participant will receive two active devices and one sham comparator in a crossover design.The cryotherapy device used consists of an opaque bag with a plastic outer cover and an aluminum interior filled with 80 grams of crushed ice. This device is applied on the skin where the optimal palpation point of the radial artery is located, where arterial puncture for blood gas analysis is usually performed to reduce skin temperature in ranges that decrease nerve conduction velocity and increase pain threshold.
  Other Names: ih1
Device: Frozen peas — Each participant will receive two active devices and one sham comparator in a crossover design. The cryotherapy device used consists of an opaque bag with a plastic outer cover and an aluminum interior filled with 80 grams of frozen peas. This device is applied on the skin where the optimal palpation point of the radial artery is located, where arterial puncture for blood gas analysis is usually performed to reduce skin temperature in ranges that decrease nerve conduction velocity and increase pain threshold.
  Other Names: ig2
Device: Room temperature gel — Each participant will receive two active devices and one sham comparator in a crossover design. The sham comparator device used consists of an opaque bag with an external plastic cover and an aluminum interior filled with 80 grams of ultrasound gel at room temperature. This device is applied on the skin where the optimal palpation point of the radial artery is located, where arterial puncture for blood gas analysis is usually performed.
  Other Names: ctrl

SUMMARY:
Low-intervention clinical trial. The thermal and hemodynamic effects of different cryotherapy devices are evaluated. This study is included in the doctoral thesis of the principal investigator.

Investigators:

Principal Investigator: Julio Alberto Mateos Arroyo (RN, MSc, PhD student) Directors: Ignacio Zaragoza García (RN, PhD), Ismael Ortuño Soriano (RN, PhD), Paloma Posada Moreno (PhD).

Setting: Faculty of Nursing, Physiotherapy and Podiatry of the Universidad Complutense de Madrid.

The three interventions to be evaluated are:

* Applying crushed ice.
* Apply frozen peas.
* Apply comparator.

Hypothesis: There are differences in the reduction of temperature, dimensions of the internal lumen of the radial artery and blood flow inside it depending on the different modalities of cryotherapy (crushed ice or bag of frozen peas) applied in the anatomical area of the wrist, point of arterial puncture for blood gas analysis.

Main objective: To analyze the effect of 3 cryotherapy devices on the radial artery area.

Secondary objectives

* To analyze the thermal behavior of the superficial tissue under study according to the cryotherapy device used.
* To analyze the differences in the radial artery caliber before and after the application of cold in the different experimental modalities under study.
* To analyze the differences in radial artery blood flow before and after the application of cold in the different experimental modalities under study.
* To identify the safety pattern of the use of the different cryotherapy devices (adverse events).

Design: Randomized controlled clinical trial. This is a crossover clinical trial in which all participants will receive all interventions and will be randomized in the order in which they receive them.

Population: Adults with a good general state of health, who specifically do not have factors that could affect their thermoregulation or vascular pathologies.

Main variables:

* Skin surface temperature.
* Radial artery size.
* Radial artery blood flow.

DETAILED DESCRIPTION:
Pain caused by arterial puncture for blood gas analysis is one of the most common problems with this procedure. The low utilization rates of effective methods by healthcare providers for pain reduction, such as subcutaneous infiltration of anesthetics, make it necessary to search for effective and simple methods. The use of cryotherapy devices has proven effective for this purpose because the decrease in temperature increases pain threshold and tolerance due to a reduction in nerve conduction velocity and inhibition of nociceptors. In order to standardize these devices, it is necessary to understand the specific thermodynamic and hemodynamic effects of these devices. At the hemodynamic level, the reduction in temperature can produce arterial vasoconstriction. This effect may decrease the palpation of the radial artery, a necessary step for the identification of the optimal point of arterial puncture. Our hypothesis is that there are differences in temperature reduction, radial artery internal lumen dimensions and blood flow inside the radial artery depending on the different cryotherapy modalities applied in the anatomical area of the wrist, the point of arterial puncture for blood gas analysis. In order to obtain an answer to this hypothesis, we will propose a randomized controlled clinical trial with a sham comparator and two active interventions: crushed ice and frozen peas. In addition, this trial has a crossover design with the aim of minimizing the differences that may arise due to individual particularities (within-group variability), and thus increase the possible effect of the interventions (between-group variability). This choice has its justification in that the application of cryotherapy, according to some studies, has a thermal reducing effect with high individual variability. In this study, adults with a good general state of health, who specifically do not have factors that could affect their thermoregulation or vascular pathologies, will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Good general health.
* Conscientious, with full cognitive and communicative capacity.
* Signed informed consent for this randomized clinical trial.

Exclusion Criteria:

* Active smoker.
* Cardiovascular disease.
* Peripheral vascular disease.
* Cyanosis of hands and fingers, Raynaud's Syndrome, Scleroderma and/or CREST Syndrome.
* Diabetes.
* Surgery, recent wounds or any type of major injury affecting the neck, shoulder girdle, upper limbs and/or hands.
* Carrier of an arterio-venous fistula.
* Lack of sensitivity to cold.
* Alcohol or caffeine intake in the last 24 hours.
* Intense physical exercise in the last 24 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Skin temperature | Prior to application of the intervention
  Surface temperature measurements will be taken at different times since the application of the interventions. The thermal camera FLIR TG267 will be used, temperature range: -25ºC to 380ºC, sensitivity <70ºC mK, resolution 160 X 120.
Skin temperature | After 5 minutes from the application of the intervention
  Surface temperature measurements will be taken at different times since the application of the interventions. The thermal camera FLIR TG267 will be used, temperature range: -25ºC to 380ºC, sensitivity <70ºC mK, resolution 160 X 120.
Skin temperature | After 10 minutes from the application of the intervention
  Surface temperature measurements will be taken at different times since the application of the interventions. The thermal camera FLIR TG267 will be used, temperature range: -25ºC to 380ºC, sensitivity <70ºC mK, resolution 160 X 120.
Skin temperature | After 15 minutes from the application of the intervention
  Surface temperature measurements will be taken at different times since the application of the interventions. The thermal camera FLIR TG267 will be used, temperature range: -25ºC to 380ºC, sensitivity <70ºC mK, resolution 160 X 120.
Skin temperature | After 20 minutes from the application of the intervention
  Surface temperature measurements will be taken at different times since the application of the interventions. The thermal camera FLIR TG267 will be used, temperature range: -25ºC to 380ºC, sensitivity <70ºC mK, resolution 160 X 120.

SECONDARY OUTCOMES:
Change in radial artery size | 0-20 minutes
  Three measurements of the anteroposterior diameter of the radial artery will be taken in the same place and plane to ensure reliability at each time point studied. Samsung HS50 ultrasound scanner with a 3-14 Hz linear probe will be used for the measurement.
Change in radial artery blood flow | 0-20 minutes
  To obtain the blood flow of the radial artery, color Doppler mode will be used to correctly identify the vessel and then the pulsed Doppler mode will be used to obtain the peak systolic low (PSV), that is, the maximum systolic velocity (VSM). Three consecutive PSV measurements will be obtained in the same place and plane to ensure reliability at each time point studied. Samsung HS50 ultrasound scanner with a 3-14 Hz linear probe will be used for the measurement.

OTHER OUTCOMES:
Discomfort | After 5 minutes from the application of the intervention
  The discomfort generated by the interventions and the comparator will be recorded 5, 10, 15 and 20 minutes after their application. An ad hoc likert-type numerical scale will be used, where 1 means no discomfort and 10 means extreme discomfort.
Discomfort | After 10 minutes from the application of the intervention
  The discomfort generated by the interventions and the comparator will be recorded 5, 10, 15 and 20 minutes after their application. An ad hoc likert-type numerical scale will be used, where 1 means no discomfort and 10 means extreme discomfort.
Discomfort | After 15 minutes from the application of the intervention
  The discomfort generated by the interventions and the comparator will be recorded 5, 10, 15 and 20 minutes after their application. An ad hoc likert-type numerical scale will be used, where 1 means no discomfort and 10 means extreme discomfort.
Discomfort | After 20 minutes from the application of the intervention
  The discomfort generated by the interventions and the comparator will be recorded 5, 10, 15 and 20 minutes after their application. An ad hoc likert-type numerical scale will be used, where 1 means no discomfort and 10 means extreme discomfort.
Adverse events | Through study completion, an average of 3 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Zaragoza García, RN, PhD, Study Director — Universidad Complutense de Madrid; Ismael Ortuño Soriano, RN, PhD, Study Director — Universidad Complutense de Madrid; Paloma Posada Moreno, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Gerencia de Atención Integrada de Talavera de la Reina, Talavera de la Reina, Toledo, Spain